CLINICAL TRIAL: NCT00446953
Title: Interest in Programming Caesarean Section at 38 Weeks of Pregnancy With Antenatal Betamethasone to Prevent Neonatal Respiratory Distress and to Avoid Emergency Caesarean Section Before Planned Date.
Brief Title: Caesarean and Corticotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3740
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neonatal Distress
Keywords: Caesarean section; Corticosteroids; Betamethasone; Neonatal distress
MeSH Terms: interventions — Betamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2x 12 mg betamethazone
  Interventions: Drug: betamethasone
- 2 (Placebo Comparator): no drugs
  Interventions: Other: placebo

INTERVENTIONS:
Drug: betamethasone — 2x12 mg betamethazone c-section at 38 weeks
  Arms: 1
Other: placebo — c-section at 39 weeks
  Arms: 2

SUMMARY:
Comparison of two randomized group :

* caesarean section planned at 38 weeks after 2 antenatal injections of 12 mg of betamethasone 48 h before.
* caesarean section planned at 39 weeks without corticosteroid.

The aim is to demonstrate that programming caesarean section at 38 weeks of pregnancy, after antenatal corticosteroid, allows to avoid caesarean section in emergency (because of a labour before 39 weeks), without increasing the neonatal respiratory distress rate.

ELIGIBILITY:
Inclusion Criteria:

* woman who needs elective caesarean section

Exclusion Criteria:

* multiple pregnancy
* toxaemia
* rhesus immunization
* fetal infection
* maternal gastro-duodenal ulcer
* mother HIV+
* prior injection of corticosteroid during the pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Neonatal respiratory distress | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Langer, MD, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (5):
- France (5):
  - Le Parc Centre pour la Mère et l'Enfant, Colmar
  - Centre Hospitalier de Haguenau, Haguenau
  - Hôpital de Hasenrain, Mulhouse
  - Cmco-Sihcus, Schiltigheim
  - Hôpital de Hautepierre, Strasbourg

REFERENCES:
- [Result] Sananes N, Koch A, Escande B, Aissi G, Fritz G, Roth E, Weil M, Bakri A, Bolender C, Meyer N, Vayssiere C, Gaudineau A, Nisand I, Favre R, Kuhn P, Langer B. Pilot randomised controlled trial comparing the risk of neonatal respiratory distress in elective caesarean section at 38 weeks' gestation following a course of corticosteroids versus caesarean at 39 weeks. Eur J Obstet Gynecol Reprod Biol. 2017 May;212:54-59. doi: 10.1016/j.ejogrb.2017.03.020. Epub 2017 Mar 10. PMID 28342389